CLINICAL TRIAL: NCT04580147
Title: A Multi-Center, Randomized, Sham-Controlled, Phase II Trial Evaluating Intravitreal Aflibercept for the Prevention of Proliferative Vitreoretinopathy Following Macula Off Rhegmatogenous Retinal Detachment Repair (The PREVENT-PVR Trial)
Brief Title: Intravitreal Aflibercept for the Prevention of Proliferative Vitreoretinopathy Following Retinal Detachment Repair
Acronym: PREVENT-PVR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: M. Ali Khan, MD (Other)
Collaborators: Southeastern Retina Associates (Unknown); Eye Associates of New Mexico (Unknown); University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, M. Ali Khan, MD, Assistant Professor, Retina Service, Wills Eye
Organization: Wills Eye (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: PREVENTPVR_V1
Record Dates: First submitted 2020-09-16; First posted 2020-10-08 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Retinal Detachment With Multiple Breaks, Unspecified Eye; Proliferative Vitreoretinopathy
MeSH Terms: conditions — Vitreoretinopathy, Proliferative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (serial IAI) (Experimental): Intravitreal aflibercept injection (2mg/0.05mL) at the conclusion of RRD repair surgery, at post-operative day 30 (+/-7 days), and at post-operative day 60 (+/-7 days)
  Interventions: Drug: Intravitreal aflibercept injection
- Control (Sham Comparator): Patients enrolled in the control group will undergo a sham procedure at post-operative day 30 (+/-7 days) and at post-operative day 60 (+/-7 days)
  Interventions: Other: Sham control

INTERVENTIONS:
Drug: Intravitreal aflibercept injection — Intravitreal aflibercept injection (2mg/0.05mL) at the conclusion of RRD repair surgery, at post-operative day 30 (+/-7 days), and at post-operative day 60 (+/-7 days)
  Other Names: Intravitreal Eylea injection
  Arms: Intervention (serial IAI)
Other: Sham control — Sham procedure at post-operative day 30 (+/-7 days), and at post-operative day 60 (+/-7 days)
  Arms: Control

SUMMARY:
The primary objective of the study is to determine if serial intravitreal aflibercept injections (IAI) improve the single surgery anatomic success rate following surgical repair of primary, macula involving rhegmatogenous retinal detachment (RRD) deemed at high risk for proliferative vitreoretinopathy (PVR). Preclinical work has revealed that competitive inhibition of platelet derived growth factor (PDGF) by vascular endothelial growth factor (VEGF) potentiates a pathologic, sustained activation of PDGF receptors that is critical to the progression of experimental PVR. VEGF blockade would mitigate this pathologic activation.

DETAILED DESCRIPTION:
The objective of this study is to determine if serial intravitreal aflibercept injections (IAI) improve single surgery anatomic success rate and reduce development of clinically apparent proliferative vitreoretinopathy (PVR) following surgical repair of primary, macula involving rhegmatogenous retinal detachment (RRD).

This will be a randomized clinical trial, with participant enrollment lasting ~120 days. 150 eyes will be randomized 1:1 to intervention (serial IAI) versus sham control (standard of care). Adult eyes with macula involving primary RRD deemed at high risk for PVR development as determined by pre-specified clinical features are eligible for enrollment.

The study, Aflibercept group will receive intravitreal aflibercept injection (2mg/0.05mL) at the conclusion of RRD repair surgery, at post-operative day 30 (plus/minus 7 days), and at post-operative day 60 (plus/minus 7 days). Patients enrolled in the control group will undergo a sham procedure at post-operative day 30 (plus/minus 7 days) and at post-operative day 60 (plus/minus 7 days).

The primary outcome will be single surgery anatomic success (retinal re-attachment) rate. Additional outcomes will include: systemic and ocular safety of IAI in setting of RRD; epiretinal membrane formation; presence of grade C PVR or worse; post-operative complication profile; OCT-measured central macular thickness; change from baseline in visual acuity (Snellen) wearing habitual correction.

All eyes will undergo pars plana vitrectomy with or without scleral buckling and gas tamponade. Post-operative exams (slit lamp biomicroscopy and indirect ophthalmoscopy) will include the following time-points: Day 30, Day 60, Day 90, Day 120. All time points will have a window of plus/minus 7 days, except the Day 120 visit which will be a window of plus/minus 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Carry a diagnosis of a macula involving ("macula off") primary RRD at high risk for PVR development. Specifically, the enrolled eye must include at least 1 but no more than 3 high risk features, which are designated as follows: multiple retinal breaks (>3); detachments involving two or more quadrants of the retina; duration of detachment > 3 weeks; vitreous hemorrhage; and choroidal detachment.
2. Consent to surgical repair utilizing pars plana vitrectomy with or without scleral buckling and C3F8 gas tamponade
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent
5. Able to understand and complete study-related questionnaires

Exclusion Criteria:

1. Age <18 years
2. Presence of PVR grade B or worse (as defined by the revised Retina Society PVR classification system) at time of surgical repair
3. Method of primary RRD repair is primary laser demarcation, primary cryotherapy, pneumatic retinopexy, or scleral buckling procedure alone.
4. Primary use of silicone oil or retinectomy during surgical repair (if silicone oil and/or a retinectomy is used intraoperatively, a prior enrolled patient will be disqualified from the study)
5. Prior incisional ocular surgery other than cataract extraction
6. History of or concurrent ruptured globe, intraocular foreign body, diabetic retinopathy, retinal vein occlusion, exudative age-related macular degeneration, macular hole, epiretinal membrane, sickle cell disease, uveitis or intraocular infectious disease
7. Treatment with intravitreal or systemic anti-VEGF pharmacotherapy in the prior 6 months.
8. Pregnant or breastfeeding women
9. Sexually active women of childbearing potential* who are unwilling to practice adequate contraception prior to start of the first treatment, during the study, and for at least 3 months after the last dose. Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Single surgery anatomic success (retinal re-attachment) rate | 4 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed on ophthalmic examination at all time points | 4 months
  Adverse events of interest include endophthalmitis, intraocular inflammation, or retinal tear/detachment.
The number of participants with an epiretinal membrane as assessed on ocular examination or optical coherence tomography imaging | 4 months
  Epiretinal membrane is defined as preretinal membrane overlying the macula.
The number of participants with evidence of grade C proliferative vitreoretinopathy (PVR) on retinal examination. Presence of grade C PVR or worse | 4 months
  PVR Grade C is defined by preretinal or subretinal retinal membrane, including a retinal star fold
Change from baseline in visual acuity (Snellen) wearing habitual correction. | 4 months
  Visual acuity will be measured using a typical Snellen chart.
OCT-measured central subfield thickness | 4 months
  Automated or manual central subfield thickness will be measured using the optical coherence tomography software.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Khan, M, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No